CLINICAL TRIAL: NCT05697367
Title: Swiss Childhood Health and Nutrition Survey 2023
Acronym: CHildHNS23
Status: Completed | Type: Observational
Sponsor: Isabelle Herter-Aeberli (Other)
Responsible Party: Sponsor-Investigator, Isabelle Herter-Aeberli, Senior Scientist, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Other Study IDs: CHildHNS23
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will repeat previous studies done in 2002, 2007 2012 and 2017/18, in order to monitor the trend in the prevalence of overweight and obesity in 6-12 year old children in Switzerland over the entire period. Furthermore, additional risk factors will be assessed for the later development of NCD using a questionnaire comparable to the one used in 2017/18.

DETAILED DESCRIPTION:
A total of ca. 2500 children will be recruited throughout Switzerland and their height, weight, waist circumference as well as percentage body fat will be measured. In addition, children will be asked to complete a questionnaire on some aspects of their diet, physical activity, health and socioeconomic background. Data will be compared to previous surveys conducted since 2002 to monitor trends in overweight and obesity prevalence in Switzerland. The results from the questionnaire will be used to investigate risk factors for obesity and the later development of NCDs.

ELIGIBILITY:
Inclusion Criteria:

* age between 6 and 12 years

Exclusion Criteria:

* none

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: School aged children living in Switzerland
Sampling Method: Probability Sample
Enrollment: 1245 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Prevalence of overweight and obesity | baseline
  Based on weight and height measurements BMI-zscores will be calculated for the classification into the different weight status groups.

SECONDARY OUTCOMES:
waist circumference | baseline
  waist circumference in cm
percent body fat | baseline
  percent body fat as calculated from 4 skinfold thickness measures
physical activity | baseline
  Assessed using a questionnaire as hours per week
Nutrition | baseline
  Assessed using a food frequency questionnaire (never to several times a week)
General health | baseline
  Assessed using a questionnaire
Parental education | baseline
  Assessed using a questionnaire on a 5 item scale ranging from obligatory schooling (lowest rating) to university degree (highest rating)
Country of birth | baseline
  Assessed in a questionnaire

OTHER OUTCOMES:
Age | baseline
  Assessed using a questionnaire, reported by parents
Sex | baseline
  Assessed using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Herter-Aeberli, PhD, Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
On request, and upon approval, anonymized data can be made available to other researchers.